CLINICAL TRIAL: NCT05480969
Title: The Effect of a Nurse-led Educational Intervention on Self-management and Prognosis of Patients With Heart Failure
Brief Title: Nurse-led Educational Intervention on Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Maria Thodi, Registered Nurse, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 28/18-01-2019
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Heart failure management programmes; Nurse-led educational interventions; Self-care; Health-related quality of life; Caregiver outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): Heart failure educational sessions will be provided by the heart failure-trained nurse to patients and caregivers. These will be delivered through a combination of home visits and telephone calls performed at regular time intervals for a total period of 6 months.
  Interventions: Other: Heart failure educational intervention
- Intervention group 2 (Experimental): Heart failure educational sessions will be provided by the heart failure-trained nurse to patients and caregivers. These will be delivered through telephone calls performed at regular time intervals for a total period of 6 months.
  Interventions: Other: Heart failure educational intervention
- Control group (No Intervention): Control patients and caregivers will receive usual care for heart failure.

INTERVENTIONS:
Other: Heart failure educational intervention — Educational intervention constitutes of a face-to-face session delivered before hospital discharge and outpatient sessions on regular intervals for a total of 6 months. Outpatient sessions in Intervention group 1 constitute of two home-based sessions on months 1 and 3, combined with weekly telephone calls during month 1 and bi-weekly calls during months 2-6. Outpatient sessions in Intervention group-2 constitute of weekly telephone sessions during month 1 and bi-weekly calls during months 2-6. The pre-discharge session will address self-monitoring and health awareness. Education will be provided by in-person discussion and through printed supporting material. Caregiver education will include understanding heart failure and advice on how to support their patient, manage their own health and well-being and how to get help when needed. During outpatient sessions, repeat education will be done and evaluation of implementation of self-care activities.
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
A randomized controlled study to examine the effect of a nurse-led, home/telephone or telephone-only educational intervention on outcomes of heart failure patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or women aged ≥18 years old.
* Hospitalized for new-onset or decompensated chronic heart failure.

Exclusion Criteria:

* Any severe neuromuscular disease or other disability or mobility problems that preclude performance of six-minute walk test.
* Any severe cognitive dysfunction or psychiatric disease that limit ability to receive education.
* Patients unable to be contacted by phone or other means.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change in the Clinical Summary Score from baseline to month 6 by Kansas City Cardiomyopathy Questionnaire (KCCQ) Greek version | Baseline, 6 months

SECONDARY OUTCOMES:
Change in the Self-Care of Heart Failure Index (SCHFI) (Greek version) from baseline to month 6 | Baseline, month 6
Change in the European Heart Failure Self-care Behavior Scale (EHFScBS-9) (Greek version) from baseline to month 6 | Baseline, month 6
Change in the Dutch Heart Failure Knowledge Scale Greek version from baseline to month 6 | Baseline, month 6
Change in the Self-rating Depression Scale-SDS (Greek version) from baseline to month 6 | Baseline, month 6
Change in the Mini Mental State Examination (MMSE) (Greek version) from baseline to month 6 | Baseline, month 6
Change in exercise capacity (6 minute walking test - 6MWT) from baseline to month 6 | Baseline, month 6
Change in plasma levels of N-terminal pro-brain natriuretic peptide (NT-proBNP) from baseline to month 6 | Baseline, month 6
Time to the first occurrence of a composite of all-cause death or heart failure hospitalization | Time from randomization to first occurrence (up to 6 months)
Change in the Caregiver Guilt Questionnaire (CGQ) (Greek version) from baseline to month 6 | Baseline, month 6
Change of the Heart Failure-Caregiver Questionnaire (HF-CQ) (Greek version) from baseline to month 6 | Baseline, month 6
Change in the EuroQol Health-Related Quality of Life Questionnaire EQ-5D three-level version (EQ-5D-3L) (Greek version) from baseline to month 6 | Baseline, month 6

CONTACTS AND LOCATIONS:
Overall Officials: Gerasimos Filippatos, Professor, Study Chair — 2nd Department of Cardiology, Attikon University Hospital
Locations (1):
- Attikon University Hospital, Chaïdári, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thodi M, Bistola V, Lambrinou E, Keramida K, Nikolopoulos P, Parissis J, Farmakis D, Filippatos G. A randomized trial of a nurse-led educational intervention in patients with heart failure and their caregivers: impact on caregiver outcomes. Eur J Cardiovasc Nurs. 2023 Oct 19;22(7):709-718. doi: 10.1093/eurjcn/zvac118. PMID 36510826